CLINICAL TRIAL: NCT02580383
Title: Effect of the Multifidus Muscle Twitch on the Long Term Effect of Radiofrequency Lumbar Medial Branch Neurotomy
Brief Title: Multifidus Muscle Twitch on the Prognosis of Lumbar Medial Branch RF
Status: Completed | Type: Observational
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Dr. Koh, Jae Chul, MD, Clinical fellow, Severance Hospital
Other Study IDs: 2015-0385-001
Record Dates: First submitted 2015-10-18; First posted 2015-10-20 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Facet Joint Syndrome
Keywords: Radiofrequency ablation; RF-MB; Lumbar RF; Facet joint syndrome; Multifidus twitching; Sensory stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group none: According to the adequacy of RF needle position while performing radiofrequency neurotomy of lumbar medial branch.
  When both needles were positioned inadequately for a facet joint.
  Interventions: Procedure: Radiofrequency neurotomy of lumbar medial branch
- Group partial: According to the adequacy of RF needle position while performing radiofrequency neurotomy of lumbar medial branch.
  when one of the needles for a facet joint medial branch was placed inadequately.
  Interventions: Procedure: Radiofrequency neurotomy of lumbar medial branch
- Group complete: According to the adequacy of RF needle position while performing radiofrequency neurotomy of lumbar medial branch.
  When all needles were placed adequately.'
  Interventions: Procedure: Radiofrequency neurotomy of lumbar medial branch

INTERVENTIONS:
Procedure: Radiofrequency neurotomy of lumbar medial branch — In above L5, The RF needle was placed to contact with bone as close as possible to the course of the target nerve in parallel. For L5 dorsal rami ablation, the needle was positioned in the groove between the S1 articular process and sacral ala. At each level, the electrodes were adjusted to optimize sensory stimulation at a frequency of 50 Hz and maximize multifidus contraction at 2 Hz. A 75 second 80°C lesion was made using an RF generator.
  Other Names: Lumbar RF neurotomy

SUMMARY:
The investigators collected data and chart from the patients who were diagnosed facet joint syndrome and underwent lumbar RF medial branch neurotomy between January 2009 and June 2014.

RF was performed using sensory stimulation and multifidus twitching to confirm the position of RF needle. The patients wil be grouped according to the adequacy of RF needle position while performing RF medial branch neurotomy ('complete' when all needles were placed adequately, 'partial' when one of the needles for a facet joint medial branch was placed inadequately, 'none' when there were both needles positioned inadequately for a facet joint) The relationship between the long term effect of RF neurotomy (longer than 6 months) and the groups will be analyzed.

DETAILED DESCRIPTION:
Facet joint syndrome has been described as a common cause of lumbar back pain. To achieve prolonged therapeutic effect in patients with lumbar facet joint syndrome, radiofrequency (RF) medial branch neurotomy is commonly performed. When performing RF neurotomy, needle placement in correct position is very important. For this reason, identification of sensory stimulation and multifidus muscle twitching by using the electrode have been commonly performed. However, there were no previous reports regarding relationship between prognosis of RF neurotomy and multifidus muscle twitching in combination of sensory stimulation. The purpose of this study was to evaluate the prognostic value of multifidus twitching when sensory stimulation was achieved while performing RF needle neurotomy in patients with lumbar facet syndrome.

The investigators have collected data and chart from the patients who were diagnosed facet joint syndrome and underwent lumbar RF medial branch neurotomy between January 2009 and June 2014.

RF was performed using sensory stimulation and multifidus twitching to confirm the position of RF needle. When numeric pain intensity score decreased less than half of the initial pain score, the procedure was regarded as effective and the duration was followed and recorded for each patients.

When multifidus twitching was observed in a voltage less than 1.0 to 2.0 times of the sensory stimulation (≤ 0.5V), the positioning of the RF needle will be regarded as adequate. The most appropriate cutoff value will be determined by univariate analysis. The patients will be grouped according to the adequacy of RF needle position while performing RF medial branch neurotomy ('complete' when all needles were placed adequately, 'partial' when one of the needles for a facet joint medial branch was placed inadequately, 'none' when there were both needles positioned inadequately for a facet joint) The relationship between the long term effect of RF neurotomy (longer than 6 months) and the groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All the patients who were diagnosed facet joint syndrome and underwent lumbar RF medial branch neurotomy between January 2009 and June 2014.

Exclusion Criteria:

* absence of 12-month follow-up data, the patients who underwent RF medial branch neurotomy on bilateral side or the patients who underwent surgery or other interventional procedures that might affect pain derived from lumbar facet joint during the follow-up period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who had lumbar back pain in Gangnam Severance hospital, Seoul, Republic of Korea.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Long term effective duration | 1 years
  Duration of pain score less than half of initial pain score

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Woo Lee, MD, PhD, Study Chair — Department of Anesthesiology and Pain medicine, Gangnam Severance Hospital, Seoul, Korea
Locations (1):
- Gangnam Severance Hospital, Seoul, Gangnam-gu, South Korea

REFERENCES:
- [Background] Cohen SP, Strassels SA, Kurihara C, Griffith SR, Goff B, Guthmiller K, Hoang HT, Morlando B, Nguyen C. Establishing an optimal "cutoff" threshold for diagnostic lumbar facet blocks: a prospective correlational study. Clin J Pain. 2013 May;29(5):382-91. doi: 10.1097/AJP.0b013e31825f53bf. PMID 23023310
- [Background] Cohen SP, Strassels SA, Kurihara C, Lesnick IK, Hanling SR, Griffith SR, Buckenmaier CC 3rd, Nguyen C. Does sensory stimulation threshold affect lumbar facet radiofrequency denervation outcomes? A prospective clinical correlational study. Anesth Analg. 2011 Nov;113(5):1233-41. doi: 10.1213/ANE.0b013e31822dd379. Epub 2011 Sep 14. PMID 21918166